CLINICAL TRIAL: NCT01532102
Title: A Double-blind, Placebo Controlled, Randomized, Phase IIa Study to Assess the Safety, Tolerability, Efficacy, and Pharmacokinetics of Repeated Topical Applications Over 42 Days of AP611074 5% Gel in Condyloma Patients
Brief Title: Safety and Efficacy Study of Topical AP611074 Gel to Treat Genital Warts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anaconda Pharma (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP611074.CT3; 2011-003760-80 (EudraCT Number)
Record Dates: First submitted 2012-01-12; First posted 2012-02-14 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Anogenital Warts; Condylomata Acuminata; Human Papillomavirus Infection
Keywords: Genital warts; Anogenital warts; HPV; Human papillomavirus; Antiviral
MeSH Terms: conditions — Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AP611074 5% gel (Experimental): Twice daily application of 100 mg dose of AP611074 5% gel for 41 days followed by a single morning application on Day 42
  Interventions: Drug: AP611074
- Placebo gel (Placebo Comparator): Twice daily application of 100 mg dose of placebo gel for 41 days followed by a single morning application on Day 42
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP611074
  Other Names: HPV antiviral; Anticondyloma drug
  Arms: AP611074 5% gel
Drug: Placebo — Placebo gel manufactured to appear identical to AP611074 5% gel
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of the topical application of AP611074 5% gel during 6 weeks on ano-genital warts caused by human papillomavirus (HPV).

DETAILED DESCRIPTION:
Genital warts (GW; also called condylomas or condylomata acuminata) are lesions caused by infection of Human papillomavirus (HPV)(specifically HPV-6 or HPV-11 types, found in > 95% of lesions). GW are sexually transmitted and affect about 1% of the sexually active population. GW represent a distressful condition for social and sexual life, especially in the cases of external condylomas. No HPV-specific antiviral treatment exists to date, and all existing therapies (either surgical or drug) have limited efficacy, with a significant level of GW recurrences and are associated with local skin reactions. AP611074 is a synthetic new chemical entity that is a potent and selective inhibitor of the interaction between two viral proteins from HPV6 and HPV11, an interaction that is a necessary step for HPV DNA replication and thus viral production. AP611074 is the "first in class" specific HPV antiviral described to treat condyloma caused by HPV infection.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patient aged between 18 and 55 years.
* External condylomas, 1-15 lesions, non-confluent and individually isolated.
* Lesions must not be internal (ie, they must not penetrate the urethral meatus, vagina or anal canal); their visualization must be complete by patients and investigators without major facilitation maneuvers and easily documented by digital pictures.
* Lesions should have a total surface smaller than 5 cm2, and an individual surface smaller than 1 cm2; lesions should be easily measured using a "French Catheter Scale".
* Lesions to be treated should have appeared between 1-6 months before screening and patients should not have received any previous condyloma treatment since their appearance.
* For patients having previous episodes of condyloma lesions, they shouldn't have received any condyloma treatment for at least 12 months before screening.

Main Exclusion Criteria:

* Patients with any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease that, in the Investigator's judgment, prevents the patients from participating to the study.
* Patients with VIN or PIN (intraepithelial neoplasia of vulva or penis; ie, Bowenoid papulosis), or genital disease (ie, lichen sclerosus, lichen planus, lichen simplex chronicus, dermatitis, psoriasis, bullous diseases, systemic diseases with genital manifestations) requiring treatment.
* Patients with fibroepithelial polyps or scaly non-viral papillomas, seborrheic keratosis, follicular papules, syringoma, or circumscribed lymphangiomas.
* Patients whose skin condition or coloration would interfere with the observation and the follow-up of the lesions during the study.
* Patients for whom a proper follow-up of the lesions during the study will not be possible, because of hair growth in the treatment area.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2013-05-06 (Actual); Study Completion 2013-05-06 (Actual)

PRIMARY OUTCOMES:
Complete or partial regression of anogenital warts, based on the total lesion surface before and after treatment | 6 weeks

SECONDARY OUTCOMES:
Safety and local tolerability | Up to 8 weeks
  Descriptive statistics will be calculated by comparing the number of subjects between Day 1 and Day 42 in each treatment group (active or placebo) presenting AEs, or changes in physical examination, vital signs (blood pressure and pulse rate), 12-lead ECG, clinical laboratory parameters (biochemistry, hematology, urinalysis), and local tolerability (erythema, scaling, stinging, oedema)
Pharmacokinetic evaluation | Up to 8 weeks
  Plasma concentrations of AP611074 will be measured from blood samples once weekly up to 8 weeks in all patients. Data will be summarized with descriptive statistics by nominal sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Chosidow, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (4):
- Argentina (2):
  - IADT - Instituto Argentino de Diagnostico y Tratamiento S.A., Buenos Aires
  - Hospotal Italinao de Buenos Aires - Dept of Dermatology and Gynecology, Buenos Aires
- France (2):
  - Hopital Henri Mondor-Dept of Dermatology, Créteil
  - SGS Aster, Paris